CLINICAL TRIAL: NCT05595616
Title: Comparison of Core Temperature Using Tracheal Thermometer and Pulmonary Artery Catheter in Adult Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Comparison of Temperature Using Tracheal Thermometer and Pulmonary Artery Catheter in Adult Patients Undergoing CABG
Acronym: TVP
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Park Seyeon, MD, Clinical assistant professor, Pusan National University Yangsan Hospital
Other Study IDs: 2022-09-01
Record Dates: First submitted 2022-10-19; First posted 2022-10-27 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Insertion of tracheal thermometer and pulmonary artery catheter — Endotracheal intubation of endotracheal tube with thermometer (Human Endotracheal Tube, Insung Medical Co., Korea) and insertion of Swan-Ganz catheter

SUMMARY:
In anesthesia, monitoring of core body temperature is one of important factors. Measurement of temperature using a pulmonary artery catheter is representative one of core temperature measurements. The core temperature by a pulmonary artery catheter is compared with the tracheal temperature by an endotracheal tube with thermometer. This study was designed to confirm the accuracy of the endotracheal tube thermometer.

DETAILED DESCRIPTION:
All patients undergoing general anesthesia are monitored core body temperature. Coronary artery bypass graft surgery needs general anesthesia with endotracheal intubation and insertion of pulmonary artery catheter. Using endotracheal tube with thermometer and pulmonary artery catheter, the investigators will measure tracheal temperature and pulmonary artery temperature every 5 minutes for 1 hour after induction of general anesthesia.

Standard monitoring devices (non-invasive BP, electrocardiogram, pulse oxygen saturation) are applied to participants in an operation room, and 1% propofol 1-2 mg/kg and rocuronium 0.8 mg/kg are administered intravenously for induction of general anesthesia. An endotracheal tube with thermometer (Human Endotracheal Tube, Insung Medical Co., Korea) is inserted. After inserting a 9Fr central venous catheter with a pulmonary artery catheter insertion port, core body temperature is measured by a pulmonary artery catheter (Swan-Ganz CCOmbo V, Edwards Lifesciences, Irvine, California, USA).

Tracheal temperature will be compared with pulmonary artery temperature by using Bland-Altman method.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18-year-old undergoing coronary artery bypass surgery

Exclusion Criteria:

* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over 18-year-old undergoing coronary artery bypass surgery using pulmonary artery catheter
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Comparison of tracheal temperature versus pulmonary artery temperature | Tracheal temperature and pulmonary arterial temperature are measured every 5 minutes for 1 hour after induction of general anesthesia.
  This study compares core body temperature measured by a pulmonary artery catheter and temperature measured by an endotracheal tube with a thermometer.
  Additional description> Time points or intervals are not important factors in this study. The study needs repeated measurements using method A (tracheal thermometer) and method B (pulmonary artery thermometer). Then it compares tracheal temperature with pulmonary artery temperature, and checks the agreement of method A and B.

CONTACTS AND LOCATIONS:
Overall Officials: Seyeon Park, MD, Principal Investigator — PNUYH, 20 Geumo-ro, Beomeo-ri, Mulgeumeup, 50612, Yangsan, Korea
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

REFERENCES:
- [Derived] Park S, Kim HY, Kim HJ, Jung J, Hong SH, Jung YS, Ha DH, Park DE, Yoon JU. Comparison of core temperature using tracheal thermometer and pulmonary artery catheter in adult patients undergoing coronary artery bypass graft surgery. PLoS One. 2025 Jan 2;20(1):e0314322. doi: 10.1371/journal.pone.0314322. eCollection 2025. PMID 39746099